CLINICAL TRIAL: NCT01327027
Title: Phase 2 Study of Vasopressin Effects on Human Social Communication
Brief Title: Vasopressin Effects on Human Social Communication
Acronym: AVP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bowdoin College (Other)
Collaborators: MaineHealth (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Richmond R. Thompson, Ph.D. Associated Professor, Bowdoin College
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 105,108; R01MH087721-02 (NIH)
Record Dates: First submitted 2011-03-30; First posted 2011-04-01 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Healthy
Keywords: vasopressin; antisocial; affiliation
MeSH Terms: conditions — Diabetes Insipidus; Antisocial Personality Disorder | interventions — Vasopressins; Arginine

STUDY DESIGN:
Intervention Model Description: In the work at Maine Medical, each subject received one of two doses of vasopressin (20IU or 40IU) on one test day, and placebo (sterile saline) on the other, in counterbalanced order. All subjects reported back for a 3rd day, 2-21 days after the 2nd test day, for a third test when no drug was administered.
  Because preliminary data analysis suggested the drug may have longer lasting, generalized effects on behavioral responses than anticipated, the second study done at Emory University with a single dose and in which subjects were also tested in fMRI, was changed to between-subjects design in which each subject either received placebo or 40IU on an initial test day and were then tested on a follow up test, 2-21 days later, when no drug was given.
Who Masked: Participant, Investigator
Masking Description: The Maine Medical Pharmacy prepared drug and placebo doses; when subjects were enrolled, the pharmacy randomly assigned the subject to a condition, and gave the unmarked nasal applicator to the subject, who was accompanied by the nurse/technician. Neither the subject nor the nurse/technician collecting data knw whether it was placebo or drug, nor which dose (20IU or 40IU) the subject would be receiving on the drug day.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vasopressin, Arginine, ADH (Experimental): We will test how vasopressin affects emotional responses to facial stimuli in healthy men and women.
  Interventions: Drug: Vasopressin, Arginine, ADH
- Sterile Salilne (Placebo Comparator): Sterile saline will be administered intranasally and emotional responses to facial stimuli measured.
  Interventions: Drug: Placebo; Sterile Saline

INTERVENTIONS:
Drug: Vasopressin, Arginine, ADH — Vasopressin will be dissolved in sterile saline and intranasally delivered in one of 2 doses to each subject (20IU, 40IU)
  Other Names: Arginine, ADH
  Arms: Vasopressin, Arginine, ADH
Drug: Placebo; Sterile Saline — Sterile saline will be delivered intranasally on a second test day, in counterbalanced order with vasopressin administration.
  Other Names: Sterile Saline
  Arms: Sterile Salilne

SUMMARY:
This research is being done because we wish to understand how a chemical produced in the brain, vasopressin, effects emotional social communication processes. Understanding how this system works in normal individuals may help us understand why some people, particularly those with autism and/or antisocial personality disorder, have dysfunctional social interactions.

This study will test the effects of 3 doses of arginine vasopressin, delivered intranasally, on physiological and behavioral responses to the faces of same- and other-sex individuals in healthy men and women.

DETAILED DESCRIPTION:
If you decide to participate you will sign this informed consent and Dr. Price will ask you questions about your medications, medical history, and how you are feeling on that particular day. You will be asked to complete a questionnaire regarding Childhood Trauma and a Brief Psychiatric Rating Scale. You will undergo a brief physical examination which includes an EKG (to look at your heart function), blood pressure and pulse by Dr. Daniel Price at the Maine Medical Center. You will also be asked to provide a urine sample for drug testing and, if you are a female, for pregnancy testing. Individuals with any positive results or results which indicate a need for medical intervention will be confidentially informed by Dr. Price and will not be allowed to participate in this study. Dr. Price will facilitate the transition to medical personnel if needed. Only Dr. Price will be aware of the results from the drug and pregnancy tests, and those results will not be shared with any other members of the research team, Bowdoin administrative officials, law enforcement officers, parents or anybody else.

If you meet the criteria for entry and agree to proceed you will be asked to submit a blood sample so we can analyze the DNA in one of your genes. All results from these tests will be kept strictly confidential and protected with a National Institutes of Mental Health confidentiality certificate. You will be required to report back to Maine Medical Center on three additional days which are one to two days apart. At visit one you will be randomized to receive one of two substances which you will self administer via a spray into your nose. You will self administer the nasal spray at visit one and visit two only. Visit three will not include the administration of the nasal spray. Neither you nor the person administering the testing will be aware if the nasal spray is vasopressin dissolved in sterile saline or sterile saline alone. The nasal spray will be in an applicator which will be provided to you upon your arrival at each study treatment visit. You will be instructed on how to use the nasal sprayer by a member of the study team.

At the start of each of the three study visits, surface skin electrodes will be attached to your palms and forearms to measure skin conductance and heart rate, respectively, and to your face to record muscle activity in your facial muscles. You will then be asked to view a series of facial images while baseline physiological measures are recorded. On the first and second visits 30 minutes following the self administration of the nasal spray, you will view another series of images and answer questions and a 5 ml (approximately one teaspoon) blood sample will be taken from your vein.

On the first and second visit days (when you receive the nasal spray) you will be advised to drink no more than 1 glass of fluid (approx. 8 oz) to prevent excess water retention in response to AVP, and refrain from caffeine consumption two hours before coming to the experiment. On each return visit you will be asked about any medications you may have taken since the last visit. If you have taken any new prescription medication or recreational substances you will not be able to proceed with the study. You will have your blood pressure and temperature measured at baseline, before administration of study drug (pre-dose), again at 5 minutes after study drug administration (post-dose), 20 minutes post dose and 60 minutes post dose. Although it is unlikely, if there are any changes in your blood pressure or body temperature Dr. Price will facilitate the need for any medical attention. If you are feeling well and there are no changes in your blood pressure, pulse or body temperature, you will be able to leave approximately one hour after study drug administration.

Each of the three subsequent visits will last approximately two hours.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women 21-30 years of age

Exclusion Criteria:

* individuals with high blood pressure or a history of seizures
* allergies
* heart problems
* psychiatric problems
* drug abuse
* pregnant All subjects will be given a preliminary medical and psychiatric exam as well as drug and (for women) pregnancy test

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 225 (Actual)
Dates: Start 2011-09; Primary Completion 2015-12 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Emotional Responses | 60 min
  Physiological and behavioral measures of emotional responses to faces will be measured 30-60 min after the intranasal delivery of the drug. Specifically, electromyographic responses to same- and other-sex faces of two facial muscles, the corrugator supercilli and the zygomaticus major, will be recorded with surface electrodes, as will electrodermal skin conductance responses and heart rate accelerations. Additionally, subjects will be asked to rate how approachable each face is on a scale where -3 is threatening and not approachable and 3 is friendly and approachable.

SECONDARY OUTCOMES:
Genetic contributions | 4 years
  Emotional responses to vasopressin administration will be correlated with polymorphic variation in the gene for the V1a vasopressin receptor. Specifically, the magnitude of the responses discussed above will be correlated with the length of a polymorphic microsatellite region of the V1a promter.

CONTACTS AND LOCATIONS:
Overall Officials: Richmond Thompson, Ph.D., Principal Investigator — Bowdoin College
Locations (1):
- Maine Medical Center, McGeachey Hall, OP Psych, Portland, Maine, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Price D, Burris D, Cloutier A, Thompson CB, Rilling JK, Thompson RR. Dose-Dependent and Lasting Influences of Intranasal Vasopressin on Face Processing in Men. Front Endocrinol (Lausanne). 2017 Sep 22;8:220. doi: 10.3389/fendo.2017.00220. eCollection 2017. PMID 29018407